CLINICAL TRIAL: NCT04897919
Title: Effectiveness and Safety of Artemether + Lumefantrine and Dihydroartemisinin + Piperaquine for the Treatment of Uncomplicated Malaria in Guinea-Bissau
Brief Title: Effectiveness and Safety of Artemether + Lumefantrine and Dihydroartemisinin + Piperaquine for Treating Malaria
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bandim Health Project (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Eurartesim2015
Record Dates: First submitted 2015-08-31; First posted 2021-05-24 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Malaria; Effectiveness
MeSH Terms: conditions — Malaria | interventions — Tablets; Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dihydroartemisinin-piperaquine (Experimental): First dose will be given supervised. The rest will be provided and the parents should take it at home.
  Dihydroartemisinin-piperaquine dosing as recommended by manufacturer
  Interventions: Drug: Dihydroartemisinin-piperaquine 160 mg/20 mg Oral Tablet
- artemether-lumefantrine (Active Comparator): First dose will be given supervised. The rest will be provided and the patients should take it at home.
  Artemether-lumefantrine dosing as recommended by manufacturer
  Interventions: Drug: Artemether-Lumefantrine 20 Mg-120 Mg Oral Tablet

INTERVENTIONS:
Drug: Dihydroartemisinin-piperaquine 160 mg/20 mg Oral Tablet — Dihydroartemisinin-piperaquine is given as recommended by manufacturer and compared to the Artemether-lumefantrine group.
  Other Names: Eurartesim
  Arms: dihydroartemisinin-piperaquine
Drug: Artemether-Lumefantrine 20 Mg-120 Mg Oral Tablet — Artemether-Lumefantrine is given as recommended by manufacturer
  Other Names: Coartem
  Arms: artemether-lumefantrine

SUMMARY:
Objective: to measure the effectiveness and safety of (artemether-lumefantrine) AL and (dihydroartemisinin-piperaquine) DP in patients (> 6 months) suffering from uncomplicated P. falciparum malaria.

Patients coming to Bandim Health Center will, if accepting, be randomised to study-arm. Medication will be provided and first dose given. Patients will be followed-up on day 7, 14, 28, and 42 with clinical evaluation, malaria film and filter-paper blood-sample for polumerase chain reaction (PCR) on re-appearing parasites. On day 21 and 35 a telephone-interview will be performed.

Primary out-come: adequate clinical and parasitological response rate on day 42. Secondary out-comes: safety, re-infection vs recrudescence, and haemoglobin on day 42.

DETAILED DESCRIPTION:
To objective of the study:

1. To measure the efficacy and safety of AL and DP in children for treating uncomplicated P. falciparum malaria.
2. To determine the capacity of each drug combination to protect against re-infection.
3. To differentiate recrudescence from re-infections using PCR based methods
4. To determine haemoglobin values on days 0 and 42
5. To determine genetic polymorphisms in P. falciparum causing reparasitaemia. Study design This will be an open label, randomized, non inferiority trial conducted at the Bandim Health Centre, Guinea-Bissau. Patients with uncomplicated malaria who meet study inclusion criteria will be enrolled, randomised to treatment with either AL or DP. Medication will be provided and first dose given at the health centre.

Efficacy and safety evaluation Treatment outcomes will be early treatment failure, late clinical failure, late parasitological failure or adequate clinical and parasitological response as defined by the WHO. All will be asked routinely about previous symptoms and about symptoms that have emerged since the previous follow up visit. All adverse events will be recorded in the case record forms.

100µL of blood will be collected on Whatman 3MM filter-paper using a capillary tube on day 0, 7, 14, 28,and 42 and whenever re-parasitaemia is detected. Filter-papers will be dried and then placed inside separate sealed plastic bags.

In order to differentiate recrudescence from a re-infection genotyping using sequential analysis of pf-glurp, pfmsp1 and pfmsp2 will be done. Drug concentrations will be assessed on the week prior to re-parasitaemia. Haemoglobin concentration will be determined on day 0, 3 and 42 using a haemocueTM.

ELIGIBILITY:
Inclusion Criteria:

* Mono-infection with P. falciparum detected by microscopy.
* Parasitemia of 1.000-200.000/µl asexual forms.
* Axillary temperature ≥37.5 ˚C or a history of fever within 24 hours.
* Ability to swallow oral medication.
* Ability and willingness to comply with the study protocol for the duration of the study and to comply with the study visit schedule.
* Informed consent

Exclusion Criteria:

* Signs or symptoms of severe malaria
* Presence of general danger signs in children under 5
* Presence of severe malnutrition.
* Any evidence of chronic disease or acute infection other than malaria.
* Regular medication which may interfere with antimalarial pharmacokinetics.
* History of hypersensitivity reactions or contraindications to AL, DP or quinine.
* Domicile outside the study area.

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 474 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Adequate clinical and parasitological response rate at day 42 | Day 42
  Cumulative percentages of children having successful treatment on day 42.

SECONDARY OUTCOMES:
re-infection vs recrudescence | Day 42
  Cumulative re-infection and recrudescence rates
Haemoglobin level | Day 42
  Haemoglobin measured on day 42

CONTACTS AND LOCATIONS:
Locations (1):
- Bandim Health Centre, Bissau, Bissau Codex, Guinea-Bissau